CLINICAL TRIAL: NCT00824304
Title: Long-Term Effects of Iron and Zinc Supplementation During Infancy on Cognitive Performance and Growth 8 Years Later: A Follow-Up Study
Brief Title: Long-term Effects of Iron and Zinc Supplementation During Infancy on Cognitive Performance and Growth
Acronym: FeZn_FU
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Collaborators: Nevin Scrimshaw International Nutrition Foundation (Other); Emory University (Other)
Responsible Party: Sponsor
Other Study IDs: MU 2007-121; IRB00003440
Record Dates: First submitted 2009-01-14; First posted 2009-01-16 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2009-01

CONDITIONS: Cognitive Function; Growth
Keywords: cognitive performance; growth; iron; zinc

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fe, Zn, Fe+Zn, Placebo: placebo comparator

SUMMARY:
The hypotheses of this study are:

1. Compared to children who received a placebo, children who received iron or zinc or iron and zinc combined will perform better on cognitive tests and will have better growth status at ages 8 to 10 years.
2. Compared to children who received iron or zinc alone, children who received iron and zinc combined will perform differently on cognitive tests and will have different growth status at 8 ages 8 to 10 years
3. Compared to children who had poorer iron and zinc status or poorer growth status before and after supplementation during infancy, children who had better iron and zinc status or better growth status before and after supplementation during infancy will perform better on cognitive tests and will have better growth status at ages 8 to 10 years.
4. Compared to children who have lower iron and zinc status, poorer growth status, or low animal source intake at ages 8 to 10 years, children who have higher iron and zinc status, better growth status, or high animal source intake at ages 8 to 10 years will perform better on cognitive tests and will have better growth status.

DETAILED DESCRIPTION:
Iron and zinc are important micronutrients for cognitive development and growth in children, particularly during infancy when brain development and physical growth are rapid. Iron and zinc deficiencies likely coexist in young children in poor developing countries due to high requirements for these micronutrients at this age, low consumption of animal products (which are rich sources of these nutrients) and similar problems of poor bioavailability from plant foods. One would expect that iron and zinc supplementation in infancy would be an appropriate strategy to promote long-term cognitive development and school achievement, but this has never been evaluated. We have many studies of the effects on micronutrient interventions in infancy but the benefits of these interventions have been assessed only in terms of outcomes in infancy. What are missing are studies of micronutrient interventions during the critical phase of infancy that report effects measured in school children and beyond. Only then will we begin to understand the full impact of micronutrient interventions in infancy on human function. From 1998 to 1999, a randomized, placebo controlled trial of iron and zinc supplementation was carried out in 609 4-6 month-old infants in Khon Kaen province, Thailand. Infants were randomized to four groups (zinc, iron, iron and zinc, placebo) and those supplemented received 10 mg of iron and/or 10 mg of zinc daily for 6 months. Improvements in iron and zinc status and in ponderal growth were found; no measures of cognitive development in infancy were included. We propose a follow-up study of these children at ages 8 to 10 years. From February to July 2006, we conducted a pilot study and were able to locate 584 or 96% of the sample. The children are all in school and we propose to assess schooling, cognitive performance (Wechsler test adapted to Thailand) and language and mathematical skills. In addition, data on physical growth, biochemical status, dietary intakes and socioeconomic status will be collected. We expect that knowledge from this study will be useful for properly assessing the full benefits of improving iron and zinc status in early childhood.

ELIGIBILITY:
Inclusion Criteria:

* All available children who received iron and zinc study during infancy

Exclusion Criteria:

* Neurological disorder

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All available children who received iron and zinc study during infancy
Sampling Method: Non-Probability Sample
Enrollment: 562 (Actual)
Dates: Start 2007-07; Primary Completion 2008-01 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
IQ score | Aug 2007-Jan 2008

SECONDARY OUTCOMES:
Anthropometry status | Aug 2007-Jan 2008

CONTACTS AND LOCATIONS:
Overall Officials: Tippawan Pongcharoen, M.Sc., Principal Investigator — Nutrition and Health Sciences Program, Emory University; Reynaldo Martorell, Ph.D., Principal Investigator — Hubert Department of Global Health, Emory University; Pattanee Winichagoon, Ph.D., Principal Investigator — Mahidol University
Locations (1):
- Ubonrat, Nampong, and Banphang district, Khon Kaen, Changwat Khon Kaen, Thailand

REFERENCES:
- [Derived] Pongcharoen T, DiGirolamo AM, Ramakrishnan U, Winichagoon P, Flores R, Martorell R. Long-term effects of iron and zinc supplementation during infancy on cognitive function at 9 y of age in northeast Thai children: a follow-up study. Am J Clin Nutr. 2011 Mar;93(3):636-43. doi: 10.3945/ajcn.110.002220. Epub 2011 Jan 26. PMID 21270383